CLINICAL TRIAL: NCT01789502
Title: Are Fully Covered Metal Stents Superior to Plastic Stents for Preoperative Biliary Decompression in Malignant Distal Bile Duct Obstruction?
Brief Title: Comparison Between Fully Covered Metal Stents and Plastic Stents in Preoperative Biliary Drainage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Tea Jun Song, Assistant Professor, Inje University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB-1210-034
Record Dates: First submitted 2013-02-05; First posted 2013-02-12 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Periampullary Cancer; Complications of Surgical Procedures or Medical Care; Disorder of Bile Duct Stent
Keywords: self-expandable metal stent; plastic stent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Plastic stents (Active Comparator): Plastic stents are inserted by ERCP
  Interventions: Device: Plastic stents
- Fully covered metal stents (Experimental): Fully covered metal stents are inserted by ERCP
  Interventions: Device: Fully covered metal stents

INTERVENTIONS:
Device: Fully covered metal stents — Fully covered metal stents were inserted by ERCP
  Other Names: BONASTENT, Standard Sci Tech, Seoul, Korea
  Arms: Fully covered metal stents
Device: Plastic stents — Plastic stents were inserted by ERCP
  Other Names: Biliary stents, Cook Endoscopy, Winston-Salem, NC
  Arms: Plastic stents

SUMMARY:
This study is a prospective, randomized study to compare of outcome of fully covered metal stents with that of plastic stents for preoperative biliary drainage in distal common bile duct cancer, pancreas head cancer or ampullary cancer with respect to the incidence of stent-related adverse events, the re-intervention rate, the effectiveness of biliary drainage, surgical outcomes and hospital stays.

DETAILED DESCRIPTION:
Pancreaticoduodenectomy is curative option in periampullary tumor. Preoperative endoscopic retrograde cholangiopancreatog-raphy (ERCP) is usually undertaken in patients with resectable disease to relieve biliary obstruction, which is thought to impair immune response, clotting, and other functions that impact intraoperative and postoperative outcomes. Despite conflicting data pertaining to preoperative biliary drainage, ERCP with biliary stenting has become standard practice in patients with periampullary malignancies. In a recent multicenter randomized trial, patients who underwent preoperative biliary drainage had a 74% rate of complications compared with 39% for those who directly underwent surgery without preoperative biliary drainage. In this trial, however, all patients underwent placement of plastic stents. In ERCP, self-expandable metal stent are being increasingly placed for palliation of malignant biliary obstruction. Compared with plastic stents, self-expandable metal stents have large caliber and have demonstrated longer patency duration. Even in patients with resectable malignant disease, self-expandable metal stents which are placed below the level of transection may not impair technical outcomes at surgery and can be safely removed along with the surgical specimen.

This prospective study is designed to compare the incidence of stent-related adverse events, the re-intervention rate, the effectiveness of biliary drainage, surgical outcomes and hospital stays in patients with periamupllary tumors who are undergone with self-expandable metal stents or plastic stents placement for preoperative biliary drainage

ELIGIBILITY:
Inclusion Criteria:

* Older than 20 years old of age
* Obstructive jaundice due to common bile duct cancer and pancreas head cancer, or ampullary cancer
* No evidence of distant metastases or locally advanced tumor

Exclusion Criteria:

* Unresectable stage of cancer
* Preoperative gastric operation that preclude ERCP (total gastrectomy and subtotal gastrectomy with B-II anastomosis)
* Severe gastric outlet obstruction or duodenal obstruction
* Severe comorbidity (Karnofsky<50%)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Adverse events related to the stent insertion | up to 4weeks
  Primary outcome parameter is adverse events related to the stent insertion includes post-ERCP pancreatitis, cholecystitis, cholangitis, bowel perforation or hemorrhage.

SECONDARY OUTCOMES:
Re-intervention rate | up to 4weeks
  Re-intervention is defined as endoscopic retrograde cholangiopancreatography or percutaneous transhepatic biliary drainage procedures which are required to achieve adequate preoperative biliary drainage after stent insertion.
Hospital stay | up to 1months
  Hospital stay is defined as the period between the date of stent insertion and that of discharge.
Surgical outcomes | up to 1months
  Surgical outcomes include the complete resection rate, complication rates related to surgery or the amount of transfusion during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Tae Jun Song, MD, PhD, Principal Investigator — Department of Internal Medicine, Inje University Ilsan Paik Hospital, Koyang, Korea
Locations (3):
- South Korea (3):
  - Daejun Eulji University Hospital, Daejun, Daejun
  - Inje University Ilsan Paik Hospital, Koyang, Gyeonggi-do
  - Asan Medical Center, Seoul, Seoul

REFERENCES:
- [Derived] Song TJ, Lee JH, Lee SS, Jang JW, Kim JW, Ok TJ, Oh DW, Park DH, Seo DW, Lee SK, Kim MH, Kim SC, Kim CN, Yun SC. Metal versus plastic stents for drainage of malignant biliary obstruction before primary surgical resection. Gastrointest Endosc. 2016 Nov;84(5):814-821. doi: 10.1016/j.gie.2016.04.018. Epub 2016 Apr 22. PMID 27109456